CLINICAL TRIAL: NCT06780644
Title: Comparison of Effectiveness and Safety of Triple Combination Cream of Fucinolone Acetonide 0.01%, Hydroquinone 4%, Tretinoin 0.05% with Mometasone Furoate 0.1%, Hydroquinone 4%, Tretinoin 0.05% in the Treatment of Melasma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, Sp.DVE, Subsp. D.K.E, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: triple combination cream
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A ( Triple combination Group) (Experimental): Group A, The treatment group, getting sunscreen cream in the morning and triple combination flucinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05% cream at night and facial soap that can be used in the morning and evening.
  Interventions: Drug: Triple combination cream
- Group B (Triple Combination Group) (Experimental): Group B, the treatment group, getting sunscreen cream in the morning and triple combination of mometasone furoate 0.1%, hydroquinone 4%, tretinoin 0.05%, cream at night and facial soap that can be used in the morning and evening.
  Interventions: Drug: Triple combination cream

INTERVENTIONS:
Drug: Triple combination cream — 1. Apply sunscreen SPF ≥30 in the morning on 2 knuckles
  2. Apply triple combination cream containing hydroquinone 40 mg, tretinoin 0.5 mg, and fluocinolone acetonide 0.1 mg at night all over the face except the area around the eyes, 1 fingertip unit (FTU) or 1 knuckle.
  Arms: Group A ( Triple combination Group)
Drug: Triple combination cream — 1. Apply sunscreen SPF ≥30 in the morning on 2 knuckles
  2. Apply triple combination cream containing mometasone furoate 0.1%, hydroquinone 4%, tretinoin 0.05% at night all over the face except the area around the eyes, 1 fingertip unit (FTU) or 1 knuckle
  Arms: Group B (Triple Combination Group)

SUMMARY:
This Research is a clinical study with a single-blind randomized controlled trial of evaluators. Clinical trial Randomized Controlled Trial (RCT) design that compares the use of a triple combination cream of flucinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05% with a triple cream combination of mometasone furoate 0.1%, hydroquinone 4%, tretinoin 0.05% in melasma therapy in RSCM-FKUI.

This study aims to Assess the effectiveness and safety of Triple Combination Cream of Fucinolone Acetonide 0.01%, Hydroquinone 4%, Tretinoin 0.05% with Mometasone Furoate 0.1%, Hydroquinone 4%, Tretinoin 0.05% in melasma patients

DETAILED DESCRIPTION:
Melasma is a skin pigmentation disorder characterized by macules or brownish patches on the face. Melasma is mostly found in women of productive age especially with Fitzpatrick skin type IV or V. Melasma is dominated by women, with the ratio of women to men being 9-10:1.4 Based on data from the Dermatology and Venereology polyclinic of Dr. Cipto Mangunkusumo Hospital, the proportion of melasma patient visits in 2022 was 1.17% of all new visits and all were female.

There are various treatment options for melasma which include sun protection, lightening medications, exfoliatives, antioxidants, resurfacing procedures, laser procedures, and light-based therapies. First-line treatments for melasma include sun protection and topical lightening medications. Topical brighteners that have become the gold standard of melasma therapy are triple combination creams and single hydroquinone. With 8-12 weeks of use, evidence has shown that a combination of compounds containing 4% hydroquinone, tretinoin, and steroids or triple cream produces a better therapeutic response than single hydroquinone.

Majid (2010) found that most patients (51.7%) had used mometasone-based triple-drug combination treatment beyond the recommended duration.

This research is a study using a Randomized Controlled Trial (RCT) design that compares the use of a triple combination cream of flucinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05% with a triple cream combination of mometasone furoate 0.1%, hydroquinone 4%, tretinoin 0.05% This study was single-blind randomized to investigators. Research subjects were randomized to determine the group for a triple combination cream of flucinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05% and a triple cream combination of mometasone furoate 0.1%, hydroquinone 4%, tretinoin 0.05%. Subjects will be divided into 28 people per group.

The research evaluation time is 12 weeks. The triple combination cream of flucinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05% group (A) and the triple cream combination of mometasone furoate 0.1%, hydroquinone 4%, tretinoin 0.05% group (B)

. all SP groups A, and B will undergo an initial physical examination in the form of a physical examination, clinical photos, mMASI score, MelasQOL-INA, dermoscopy, Wood's lamp, and mexameter.

Group A or B evaluation will be carried out every 4 weeks, namely weeks 0, 4, 8, 12. Subjects were given facial wash, sunscreen, and triple combination for the night Each evaluation will be checked: Physical examination , mMASI score, PtGA, mexameter examination Data is recorded in the research status which is then compiled into a master table, inputted into Ms Excel, and analyzed using SPSS for windows version 25.0. The results of the study were displayed in the form of narratives, tables, and graphs. Categorical data were presented in frequencies and percentages. Numerical data were presented as mean and standard deviation if normal data distribution was obtained or median and minimum-maximum values if abnormal data distribution was obtained.

The Pearson test is used to assess the correlation between mMASI and MELASQoL-INA scores if a normal data distribution is obtained, while the Spearman test is used if the data distribution is not normal. The test results obtained are in the form of a correlation coefficient (r) which is in the range -1 and 1. The r value which is in the range 0.1-0.3 indicates the correlation between the two variables is weak, the range 0.4-0.6 indicates a moderate correlation , a range of 0.6-0.9 indicates a strong correlation, and 1 indicates a perfect correlation. The value of statistical significance in the research is determined.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Diagnosed with melasma based on clinical and Wood's lamp examination
* 30-59 years old
* Skin type IV or V

Exclusion Criteria:

* Plan to be pregnant and breastfeeding women during the study period ( 12 weeks)
* using or have used hormonal contraception in the last 6 months, or plan to use hormonal contraception during the study period (12 weeks)
* Using topical melasma treatments such as corticosteroids, tretinoin, hydroquinone, and other skin whitening or lightening treatments in at least the last 2 weeks.
* Have used topical therapy for melasma i.e. triple combination cream for at least 3 months and showed no significant improvement.
* Using systemic therapy for melasma, e.g. antioxidants, tranexamic acid in at least the last 4 weeks.*
* History of eppeeling, laser or mechanical abrasion on the face in the last 6 months.*
* Using photosensitizer drugs such as tetracycline, phenytoin, carbamazepine, and spironolactone in at least the last 4 weeks.
* Having other skin complaints that may interfere with the evaluation of melasma such as post-inflammatory hyperpigmentation, Hori nevus, Ota nevus, pigmented contact dermatitis, and other pigmentation disorders.
* Difficulty in adherence to treatment such as long distance from home, work schedules, and busy activities.

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2025-05-26 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of Melasma Severity based on modified Melasma Severity Index (mMASI) score | re-evaluation on day 28, 56 and day 84 of therapy
  The range of values for mMASI is between 0 and 24 which can then be divided into mild melasma (0-8), moderate (8-16), and severe (16-24). improvement occurs if the mMASI score decreases by <50% from the previous visit worsening if score persists or mMASI Score Increase >50%
Change of Melasma Severity based on Patient's Tolerability Assesment (PtGA) | re-evaluation on day 84 of therapy
  one method of evaluating the response to therapy in melasma which is assessed subjectively by the patient. The response to therapy can be assessed as follows No or slight response: < 25% improvement Moderate response: 25% - 50% improvement Good response: 50% improvement - < 75% Excellent response: improvement > 75% The response is said to be good if the score is above 50% since the previous visit
Change of Melasma Severity based on Dermoscopy | re-evaluation on day 84 of therapy
  based on Dermoscopy Telangiectasis score assessment using a 5-point dermoscopy-scale: 0 = No visible capillaries. 1 = Elongated capillaries accompanied by dilation, not visible to the naked eye. 2 = Moderate telangiectasis that is beginning to be visible to the naked eye. 3 = Severe telangiectasis characterized by reduced capillary loops. 4 = Very severe telangiectasis characterized by dilatation and loss of capillary loops.
Change of Melasma Severity based on Wood's Lamp | re-evaluation on day 84 of therapy
  Epidermal Type/ Dermal Typed/ Mixed Typed
Compare Quality Of Life based on MelasQoL Score | re-evaluation on day 28, 56 and day 84 of therapy
  based on MelasQoL Score minimum score: 7 maximum score : 70
Change of Melanin Index Based on Mexameter | re-evaluation on day 28, 56 and day 84 of therapy
  improves if there is a decrease in melanin levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in melanin levels or there is a decrease of <50%
Change of Erytema Index Based on Mexameter | re-evaluation on day 28, 56 and day 84 of therapy
  improves if there is a decrease in Erytema levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in erythema levels or there is a decrease of <50%

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Central Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided